CLINICAL TRIAL: NCT06136715
Title: Massive Transfusion in Trauma Patient Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 029.TRA.2023.D
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: blood products as a part of Massive Transfusion Protocol — This data repository will serve as a means to aggregate and analyze best practices as relative to MTP in the trauma patient, with specific interest in component best practices, whole blood protocols, and electrolyte/metabolite replacement

SUMMARY:
The early use of blood products as a part of Massive Transfusion Protocol (MTP) during trauma resuscitation has been increasingly supported by providers and backed by the literature. However, the incidence of hypocalcemia during MTP has also been recorded and continues to be studied as an exacerbating factor in coagulopathy during trauma.

DETAILED DESCRIPTION:
Although initially it was thought that the coagulopathy was due to the trauma itself, studies suggest that it is worsened by the transfusion of blood as this is associated with increased hypocalcemia. The level of hypocalcemia is said to correlate with the amount of blood products transfused, but the number of units needed to produce a particular degree of hypocalcemia remains to be defined. A standardized value for hypocalcemia due to MTP has yet to be established. Establishing this value would be helpful in determining what level actually affects the rate of mortality. Some studies suggest intravenous calcium supplement should be considered during massive transfusion while others state this does not make a difference.

This data repository will serve as a means to aggregate and analyze best practices as relative to MTP in the trauma patient, with specific interest in component best practices, whole blood protocols, and electrolyte/metabolite replacement.

ELIGIBILITY:
Inclusion Criteria:

* • ≥18 years old

  * Included in the Methodist dallas medical center(MDMC) trauma registry
  * Flagged for MTP activation and/or >1unit(U) blood product recorded in the first 24 hours

Exclusion Criteria:

* • <18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ≥18 years old
  * Included in the MDMC trauma registry
  * Flagged for MTP activation and/or >1U blood product recorded in the first 24 hours
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-07-13 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
Establish a data set that will be permissive of quality improvement studies/observations specific to MTP in the trauma patient. | 5 YEARS
  This data repository will serve as a means to aggregate and analyze best practices as relative to MTP in the trauma patient, with specific interest in component best practices, whole blood protocols, and electrolyte/metabolite replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Conner McDaniel, MD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years